CLINICAL TRIAL: NCT00150956
Title: Study Into the Effects of Daily Home Hemodialysis on Hemodynamics, Neurocognitive Functions, and Quality of Life
Brief Title: Effects of Daily Home Hemodialysis on Circulation, Mental Functions, and Quality of Life
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UMC Utrecht (Other)
Collaborators: Dianet Dialysis Centers (Other); Dutch Kidney Foundation (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C98-1750; Dutch Kidney Foundation
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2005-09-08 (Estimated); Status verified 2000-10

CONDITIONS: End-Stage Renal Disease
MeSH Terms: conditions — Kidney Failure, Chronic

INTERVENTIONS:
Procedure: Daily home hemodialysis

SUMMARY:
This study was designed to discover mechanisms responsible for the decrease in (high) blood pressure after starting daily hemodialysis, as has been observed by various investigators. We hypothesized that better control of body water and sodium content and a decline in the autonomic (sympathetic) nervous system activity, increased in chronic renal failure patients, would contribute to improved blood pressure regulation.

Moreover, we studied the effects of daily hemodialysis on mental functions, like information processing and memory, in relation to the previously reported improvement in quality of life, and the effects on nutrition. We hypothesized that all would improve.

DETAILED DESCRIPTION:
Although conventional hemodialysis has faced many technical improvements in recent years, a great deal of end-stage renal disease patients, treated with this modality, have suboptimal or high blood pressure, and suffer poor quality of life. Daily hemodialysis has been reported to improve both, but the pathophysiological background is poorly understood.

Patients were studied before and after 6 months of daily (i.e.6 times a week) home hemodialysis, and again after two months of conventional (i.e. thrice weekly) hemodialysis.

We measured the effects of daily dialysis (compared with conventional dialysis) on blood pressure, cardiac output, extracellular fluid volume, plasma renin activity, sympathetic nervous system activity (through MSNA), the electroencephalogram (EEG), neurocognitive functioning (speed of information processing, memory, executive functioning, and attention), quality of life, and nutritional status

ELIGIBILITY:
Inclusion Criteria:

* End-stage renal disease patients
* Fit and motivated for home hemodialysis

Exclusion Criteria:

* Patients, who were treated with frequent dialysis (5 or 6 times a week) before
* Diabetes mellitus
* Severe comorbidity (e.g. malignancies)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12
Dates: Start 1999-04; Study Completion 2002-01

PRIMARY OUTCOMES:
Blood pressure at 6 months
Cardiac output at 6 months
Extracellular fluid volume at 6 months
Plasma renin activity at 6 months
Muscle sympathetic nerve activity (MSNA) at 6 months
Electroencephalogram (EEG) at 6 months
Neurocognitive functioning at 6 months
Quality of life at 6 months

SECONDARY OUTCOMES:
Nutritional status at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Pieter F Vos, MD, Principal Investigator — UMC Utrecht, Department of Nephrology & Hypertension
Locations (1):
- UMC Utrecht, Department of Nephrology & Hypertension, Utrecht, Netherlands

REFERENCES:
- [Background] Kooistra MP, Vos J, Koomans HA, Vos PF. Daily home haemodialysis in The Netherlands: effects on metabolic control, haemodynamics, and quality of life. Nephrol Dial Transplant. 1998 Nov;13(11):2853-60. doi: 10.1093/ndt/13.11.2853. PMID 9829490
- [Background] Vos PF, Zilch O, Kooistra MP. Clinical outcome of daily dialysis. Am J Kidney Dis. 2001 Jan;37(1 Suppl 2):S99-S102. doi: 10.1053/ajkd.2001.20761. PMID 11158871